CLINICAL TRIAL: NCT03184376
Title: Histological Improvement of Non-alcoholic Steatohepatitis With a Prebiotic: a Pilot Clinical Trial
Brief Title: Histological Improvement of NASH With Prebiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-23936
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Gut microbiota; Prebiotic; Liver biopsy; Oligofructose
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Single-blind, placebo controlled, randomized trial
Who Masked: Participant
Masking Description: Participants were blinded to the treatment allocation. Oligofructose and maltodextrin taste and look the same (white powder) and both were placed in identical foil packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Experimental): Prebiotic oligofructose (Orafti P95, Beneo-Orafti Inc., Tienen, Belgium) taken 8g orally per day for 12 weeks followed by 16g per day for 24 weeks.
  Interventions: Dietary Supplement: Prebiotic oligofructose
- Placebo (Placebo Comparator): Placebo maltodextrin (isocaloric to prebiotic) taken 3.3g orally per day for 12 weeks followed by 6.6g per day for 24 weeks.
  Interventions: Dietary Supplement: Placebo maltodextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic oligofructose — Powder format
  Arms: Prebiotic
Dietary Supplement: Placebo maltodextrin — Powder format
  Arms: Placebo

SUMMARY:
This trial will investigate the therapeutic potential of a prebiotic supplement to improve histological parameters of NASH. In a single-blind, placebo controlled, randomized pilot trial will be conduced in individuals with liver biopsy confirmed NASH (Non-alcoholic fatty liver activity score (NAS) ≥ 5). Participants will be randomized to receive oligofructose (8 g/day for 12 weeks and 16g/day for 24 weeks) or isocaloric placebo for 9 months. The primary outcome measure is the change in liver biopsy NAS score and the secondary outcomes include changes in body weight, body composition, glucose tolerance, serum lipids, inflammatory markers, and gut microbiota.

DETAILED DESCRIPTION:
Oligofructose and maltodextrin are both white powders that taste and look the same. They were both package in individual foil packets. Participants were blinded to the treatment allocation. Adherence to supplement protocol was monitored throughout the study through direct questioning and counting unused supplement packages. Participants were asked to maintain their usual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy confirmed NASH (NAS score greater than or equal to 5)
* BMI >25 kg/m2 (Caucasians)
* >23 kg/m2 (Asians)
* History of Serum ALT >1.5X upper normal limit
* No changes in lipid-lowering or diabetes medication over previous three months
* Ability to provide informed consent

Exclusion Criteria:

* alcohol consumption >20g/day (women) or >30g/day (men)
* alternate etiology for abnormal liver enzymes
* decompensated liver disease
* use of orlistat, liraglutide, prebiotic, probiotic, or antibiotic within 3 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Histological change | 9 months
  Nonalcoholic fatty liver disease activity score

SECONDARY OUTCOMES:
Body composition | 9 months
  Body lean and fat mass
Body weight | 9 months
  Body weight measurement
Glucose tolerance | 9 months
  Oral glucose tolerance test
Gut microbiota | 9 months
  Intestinal microbiota composition
Serum total cholesterol | 9 months
  Total cholesterol
Serum LDL cholesterol | 9 months
  Low-density lipoprotein cholesterol
Serum triglycerides | 9 months
  Triglycerides
Serum HDL cholesterol | 9 months
  High-density lipoprotein cholesterol
Serum IL-6 | 9 months
  Interleukin-6
Serum TNF-alpha | 9 months
  Tumor necrosis factor - alpha

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — The University of Calgary

IPD SHARING:
Plan to Share IPD: Undecided
Other researchers would need to make an individual inquiry.

REFERENCES:
- [Derived] Bomhof MR, Parnell JA, Ramay HR, Crotty P, Rioux KP, Probert CS, Jayakumar S, Raman M, Reimer RA. Histological improvement of non-alcoholic steatohepatitis with a prebiotic: a pilot clinical trial. Eur J Nutr. 2019 Jun;58(4):1735-1745. doi: 10.1007/s00394-018-1721-2. Epub 2018 May 19. PMID 29779170